CLINICAL TRIAL: NCT02236416
Title: Physical Exercise and Prevention of Cognitive Decline in Subjects at Risk of Dementia: a Randomized Controlled Trial
Brief Title: Physical Exercise for Prevention of Dementia
Acronym: EPD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Molise (Other)
Responsible Party: Principal Investigator, Alfonso Di Costanzo, MD, MD, Professor of Neurology, University of Molise
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 21933_III/11
Record Dates: First submitted 2014-09-03; First posted 2014-09-10 (Estimated); Last update posted 2021-07-21 (Actual); Status verified 2021-07

CONDITIONS: Memory Disorders; Mild Cognitive Impairment; Aging
Keywords: Dementia; Prevention; Physical Activity
MeSH Terms: conditions — Memory Disorders; Cognitive Dysfunction; Dementia; Motor Activity | interventions — Control Groups

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention group (Experimental): Physical exercise
  Interventions: Behavioral: Intervention group
- Control group (Other): Posture Education/Unchanged condition
  Interventions: Behavioral: Control group

INTERVENTIONS:
Behavioral: Intervention group — Supervised, multimodal physical activity including aerobic, resistance and stretching exercises
  Arms: Intervention group
Behavioral: Control group — Usual physical activity, generally consisting in long walks and/or stretching, toning and/or balance exercises, or posture education
  Arms: Control group

SUMMARY:
The principal aim of this study is to verify whether a program of supervised, multimodal physical exercise improves cognitive function and/or reduces the rate of cognitive decline in older adults

DETAILED DESCRIPTION:
Community-dwelling volunteers, recruited from social centers, were invited to an in-person assessment that included a medical history questionnaire and examination, anthropometric measurements, blood tests for cardiovascular risk, and several outcome measures. Participants meeting the inclusion criteria were divided in 3 groups (participants without subjective or objective cognitive impairment, with subjective memory complaints and with mild cognitive impairments) and randomly assigned (1:1) to an experimental group or a control group, using a list of random numbers generated by a statistical software. The list was kept in a sealed envelope and a researcher, not directly involved in the recruitment and in the evaluation of the participants, assigned the allocation numbers.

ELIGIBILITY:
Inclusion Criteria:

Age > 50 years old

Exclusion Criteria:

* Medical conditions that compromise survival or limit physical activity
* Geriatric Depression Scale-15 score of 6 or higher
* Alcohol intake > 4 units/day
* Mini- Mental State Examination < 24
* Clinical Dementia Rating score of 1 or more

Ages: 50 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1000 (Actual)
Dates: Start 2011-05; Primary Completion 2020-07 (Actual); Study Completion 2020-07 (Actual)

PRIMARY OUTCOMES:
Change of Mini Mental State Examination (MMSE) score from baseline to 48 months | Baseline and every 6-12 months, over an intervention period of 48 months
  Scale for grading cognitive function

SECONDARY OUTCOMES:
Change of neuropsychological test battery from baseline to 48 months | Baseline and every 6 -12 months, over an intervention period of 48 months
  It includes: Frontal Assessment Battery, Rey's Auditory Verbal Learning Test, Prose Memory, Stroop Color Word Interference Test, Attentive Matrices, Raven's Progressive Matrices, Trial Making Test, designs copying with and without programming models.
Change of Geriatric Depression Scale (GDS) from baseline to 48 months | Baseline and every 6 -12 months, over an intervention period of 48 months
  A self-report assessment for identifing depression in the elderly
Change of Short-form Health Survey (SF-36) from baseline to 48 months | Baseline and every 6 -12 months, over an intervention period of 48 months
  Assessment of health status
Change of Memory Complaint Questionnaire (MAC-Q) from baseline to 48 months | Baseline and every 6 -12 months, over an intervention period of 48 months
  Assessment of subjective memory complaint
Change of Physical Activity Scale for the Elderly (PASE) from baseline to 48 months | Baseline and every 6 -12 months, over an intervention period of 48 months
  Assessment of physical activity level in elderly
Change of AAHPERD (American Alliance for Health, Physical Education, Recreation and Dance) fitness test battery from baseline to 48 months | Baseline and every 6 -12 months, over an intervention period of 48 months
  Functional fitness assessment

OTHER OUTCOMES:
Change of Composite cognitive score (CCS) from baseline to 48 months | Baseline and every 6 -12 months, over an intervention period of 48 months
  It is calculated by averaging the standardized scores (Z-score) of all neuropsychological tests, for assessing the overall changes in cognitive performance.

CONTACTS AND LOCATIONS:
Overall Officials: Alfonso Di Costanzo, MD, Principal Investigator — University of Molise
Locations (1):
- Center for Research and Training in Medicine of Aging (CeRMA), Campobasso, Molise, Italy

REFERENCES:
- [Derived] Iuliano E, di Cagno A, Cristofano A, Angiolillo A, D'Aversa R, Ciccotelli S, Corbi G, Fiorilli G, Calcagno G, Di Costanzo A; EPD Study Group. Physical exercise for prevention of dementia (EPD) study: background, design and methods. BMC Public Health. 2019 May 29;19(1):659. doi: 10.1186/s12889-019-7027-3. PMID 31142290